CLINICAL TRIAL: NCT07342647
Title: Optimization of Perioperative Antibiotic Prophylaxis in Patients Allergic to Beta-lactams in the Orthopedic Surgery and Trauma Departments of the Strasbourg University Hospitals
Brief Title: Optimization of Perioperative Antibiotic Prophylaxis in Patients Allergic to Beta-lactams in the Orthopedic Surgery and Trauma Departments
Acronym: ORTHO-PEN
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Other Study IDs: 9812
Record Dates: First submitted 2026-01-06; First posted 2026-01-15 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2026-01

CONDITIONS: Beta Lactam Adverse Reaction
Keywords: Beta Lactam Adverse Reaction; Antibiotic Prophylaxis; Beta-Lactamines; Orthopedic Surgery

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
When surgery is required, a consultation with an anesthesiologist is mandatory. This preoperative consultation allows for the selection of the appropriate antibiotic prophylaxis tailored to the patient and the type of procedure. The French Society of Anesthesiology and Intensive Care (SFAR) has published recommendations on antibiotic prophylaxis for different types of surgery. During this consultation, several topics are addressed, including drug allergies. This topic plays a central role in the choice of antibiotic prophylaxis.

Ten percent of the population is labeled as allergic to beta-lactams, but only 1% actually are. Diagnosis is difficult and requires specialized teams. In response to the significant increase in patients labeled as allergic, and consequently the rise in requests to specialists, a scoring system has been developed for use by all physicians: the PEN FAST score. This score stratifies the risk of a true penicillin allergy and guides the selection of delabeling strategies. The test aims to eliminate the need for skin prick tests and allows for the direct reintroduction of the drug when the score is below 3. It is based on five questions. Each question is assigned a point value, which is used to calculate a score and thus an estimated risk.

The primary objective of this study is to improve the management of patients allergic to beta-lactams in orthopedic and trauma surgery by ensuring optimal and appropriate intraoperative antibiotic prophylaxis.

ELIGIBILITY:
Inclusion Criteria:

* Adult patient (≥ 18 years old)
* Patient operated on at Strasbourg University Hospital between January 1, 2023, and December 31, 2023, for total knee, shoulder, or hip replacement.
* Patients who underwent surgery at Strasbourg University Hospital between March 1, 2025, and July 31, 2025, involving surgery requiring intraoperative antibiotic prophylaxis.

Exclusion Criteria:

* Patients with a surgical indication without the use of implants.
* Patients with a surgical indication without antibiotic prophylaxis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients treated at Strasbourg University Hospital
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2025-07-11 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2026-07-11 (Estimated)

PRIMARY OUTCOMES:
Evolution of the rate of compliant prescriptions for intraoperative antibiotic prophylaxis in patients declared allergic to beta-lactams | Up to 12 months
  Rate trend:
  Trend refers to how this rate changes over time. We want to see if:
  * The rate increases: therefore, there are more correct prescriptions
  * The rate remains stable
  * The rate decreases: therefore, there are more prescription errors.

CONTACTS AND LOCATIONS:
Locations (1):
- Service de Pharmacie - Stérilisation - CHU de Strasbourg - France, Strasbourg, France